CLINICAL TRIAL: NCT04144361
Title: Outcomes of Standard Sleeve Pouch Versus Relatively Wide Pouch With Plication
Brief Title: Standard Sleeve Pouch Versus Relatively Wide Pouch With Plication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor and consultant of general surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fac,med 19.32
Record Dates: First submitted 2019-10-20; First posted 2019-10-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Morbid
Keywords: post sleeve gastrectomy leak; post sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeve without plication (Experimental): sleeve gastrectomy on bougie 36 without plication
  Interventions: Procedure: sleeve without plication
- sleeve with plication (Active Comparator): sleeve gastrectomy on bougie 42 without plication
  Interventions: Procedure: sleeve with plication

INTERVENTIONS:
Procedure: sleeve with plication — sleeve with plication
  Arms: sleeve with plication
Procedure: sleeve without plication — sleeve without plication
  Arms: sleeve without plication

SUMMARY:
three hundred morbidly obese patients candidate for sleeve gastrectomy will divided into equal two groups, group A : will operated by standard sleeve gastrectomy on bougie 36 without plication of stable line and group B: will operated by sleeve gastrectomy on bougie 42 with plication of stable line. the aim is to test the effect of pilcation on the incidence of leaks and bleeding

DETAILED DESCRIPTION:
three hundred morbidly obese patients candidate for sleeve gastrectomy will divided into equal two groups, group A : will operated by standard sleeve gastrectomy on bougie 36 without plication of stable line and group B: will operated by sleeve gastrectomy on bougie 42 with plication of stable line. the primary outcomes is the incidence of leaks and bleeding which is the main nightmare of sleeve gastrectomy, secondary outcome operative time, weight loss and metabolic effect

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative stable line bleeding | 2-24 hours
  early postoperative bleeding from stable line
the incidence of stable line leakage | 1-30 days
  leak from stable line

CONTACTS AND LOCATIONS:
Overall Officials: alaa M Sewefy, Principal Investigator — Minia University
Locations (2):
- Egypt (2):
  - Faculty of medicine, Minya
  - Minya university hospital, Minya